CLINICAL TRIAL: NCT01685372
Title: Immunogenicity and Efficacy of High-dose Trivalent Inactivated Seasonal Influenza Vaccine (Fluzone High Dose) in Immunocompromised Children and Young Adults.
Brief Title: Immunogenicity of Fluzone High Dose in Immunocompromised Children and Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12-0829
Record Dates: First submitted 2012-08-27; First posted 2012-09-14 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Solid Organ Transplant Recipient (Liver, Kidney, Heart); Rheumatologic Disorder; Human Immunodeficiency Virus (HIV); Bone Marrow Transplant (BMT); Dialysis
MeSH Terms: conditions — Collagen Diseases; Acquired Immunodeficiency Syndrome | interventions — Fluzone High-Dose; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluzone High Dose (Experimental): Fluzone High Dose 0.5 mL intramuscularly (IM) given once
  Interventions: Biological: Fluzone High Dose
- Fluzone (Active Comparator): Fluzone 0.5mL IM given once
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluzone High Dose — A single-dose of high-dose influenza vaccine will be administered to subjects randomized to this arm
  Other Names: high-dose influenza vaccine; influenza vaccine
  Arms: Fluzone High Dose
Biological: Fluzone — A single-dose of standard-dose influenza vaccine will be administered to subjects randomized to this arm
  Other Names: influenza vaccine
  Arms: Fluzone

SUMMARY:
The purpose of this study is to determine whether Fluzone High Dose increases the immune response to the influenza antigens contained in the vaccine compared to standard-dose Fluzone in immunocompromised children and young adults. Safety and efficacy data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years and ≤ 35 years
* Receiving influenza vaccination in Children's Hospital Colorado (CHC) clinic as part of routine clinical care
* Only supposed to receive one dose of influenza vaccine
* Rheumatology patients: must be on some type of immunosuppressive or immunomodulatory medication at the time of immunization and considered at least moderately immunosuppressed in the opinion of the primary rheumatologist. Basic guidelines for rheumatology patients: (1) Any patient receiving monoclonal antibody therapy (i.e., infliximab, etanercept, tocilizumab, anakinra) must also be taking another immunosuppressive/immunomodulatory medication; (2) Patients taking steroids as monotherapy must be on a dose of ≥ 2mg/kg/day OR ≥ 20mg/day; (3) Patients on combination therapy where the dose of a single drug may not be very high, but the combination is considered moderately or severely immunosuppressive will be eligible.
* Bone Marrow Transplant patients: all patients in clinic eligible
* Oncology patients: must be on some type of chemotherapy
* Hemodialysis patients: must be on dialysis
* Child Health Immunodeficiency Program (CHIP) patients: must have a known diagnosis of HIV
* Solid Organ Transplant patients: post-transplant, influenza vaccine recommended by primary transplant physician

Exclusion Criteria:

* Rheumatology patients: if receiving any of the monoclonal antibodies, etanercept, infliximab, adalimumab, tocilizumab, atlizumab, or anakinra, must also be taking at least one other immunosuppressive/immunomodulatory medication
* Unable to come for scheduled follow-up appointments
* History of anaphylaxis reaction to influenza vaccination in the past
* Severe allergic reaction to any component of the vaccine, including egg protein, or after previous dose of any influenza vaccine
* History of Guillain-Barre syndrome ever in the past in the subject or in a parent or a sibling of the subject
* Allergy to latex
* Intravenous immuneglobulin (IVIG) within in 4 weeks preceding any blood draw
* Receiving an investigational agent as part of another study or other medical treatment (investigational = not-FDA approved for any indication)
* Subject not enrolled in other studies that prohibit him/her from enrolling in this study
* Blood draw contraindicated
* Pregnancy
* Breastfeeding
* Received a polysaccharide vaccine (pneumovax) w/in 3 weeks of the vaccination
* Absolute neutrophil count (ANC) < 500/uL at the time of vaccination or could potentially have ANC 500/uL during the 5 days after vaccination
* Platelet count < 50,000/uL at the time of vaccination
* If a subject has a temperature ≥ 100.4°F at the time of enrollment, then the subject must choose to not enroll or delay immunization until afebrile.
* Receiving influenza vaccination past December 15 of influenza season.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Curtis, MD, MPH, Principal Investigator — Children's Hospital Colorado, University of Colorado Denver School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at the end of the study. Data management at the close of the study will occur according to IRB and FDA regulations.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited over two influenza seasons, 2013-2014 and 2014-2015. Subjects were recruited from the Dialysis unit and Rheumatology clinic in 2013-2014 by referral from clinicians. Subjects were recruited by mailed letter to Solid Organ Transplant recipients in 2014-2015.
Pre-assignment Details: In 2013-2014, 4 subjects chose not to enroll after learning more about the study. In 2014-2015, 2 subjects chose not to enroll after learning about the study. All potential subjects met pre-screening criteria. No subjects were excluded from the study by study personnel.
Groups:
- Fluzone High Dose: A single-dose of high-dose influenza vaccine was administered to subjects randomized to this arm at T1
- Fluzone Standard Dose: A single-dose of standard-dose influenza vaccine was administered to subjects randomized to this arm at T1
Period: Timepoint 1 (T1): Vaccine,1st Blood Draw
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Timepoint 2 (T2): 2nd Blood Draw
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Timepoint 3 (T3): 3rd Blood Draw
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Started | 7 | 9
Completed | 4 | 5
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Fluzone Standard Dose: Fluzone 0.5mL IM given once
  Fluzone: A single-dose of standard-dose influenza vaccine will be administered to subjects randomized to this arm
- Total: Total of all reporting groups
Arm/Group | Fluzone High Dose | Fluzone Standard Dose | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Median (Full Range); unit: years] | 15 [9 to 18] | 15 [10 to 23] | 15 [9 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Cohort [Count of Participants; unit: Participants]
  Dialysis | 3 | 4 | 7
  Solid organ transplant | 4 | 4 | 8
  Rheumatoloty | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Influenza and Influenza-Like-Illness Reported in High Dose and Standard Dose Vaccination Groups
Description: Gathered data on influenza and influenza-like-illness during the influenza season for which the subject was vaccinated. Reported numbers of episodes of PCR-diagnosed influenza and rates of reported Influenza-Like-Illness (ILI) from Questionnaire #2 and also that were obtained from medical records. Data were categorized by the following:
  1. Polymerase chain reaction (PCR)-proven diagnosis of influenza performed at Children's Hospital Colorado (CHC)
  2. Diagnosis of influenza by non-PCR rapid-influenza test
  3. Diagnosis of ILI (from questionnaire #2). [Centers for Disease Control (CDC) definition of ILI: Fever ≥ 100°F AND cough or sore throat in the absence of another known cause other than influenza for the illness.]
Time Frame: up to 10 months after vaccination
Population: Row 1: Number of influenza episodes diagnosed by PCR Row 2: Number of influenza episodes diagnosed by non-PCR rapid test Row 3: Number of influenza-like-illness (ILI) episodes reported by participants from the time of vaccination through June of the following year (end of flu season).
Measure: Number; unit: episodes of illness
Groups:
- Fluzone Standard Dose: Fluzone: A single-dose of standard-dose influenza vaccine will be administered to subjects randomized to this arm
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
episodes of illness
  Row 1: Number of Influenza diagnosed by PCR | 1 | 1
  Row 2: # of Influenza diagnosis by non-PCR test | 0 | 0
  Row 3: Number of Influenza-like-illness | 2 | 8

2. Primary Outcome: Number of Subjects Seroprotected at Timepoint 2 in High Dose and Standard Dose Vaccination Groups
Description: Measure hemagglutinin inhibition (HAI) on blood samples #2 for all subjects, which is the sample drawn at the "peak" of the immune response. Compare number of subjects who are seroprotected (reaching HAI ≥ 1:40) between the high-dose and standard-dose recipients..
Time Frame: blood draw at 10-45 days post-vaccination
Population: All participants had blood drawn before vaccination and at timepoint 2. The influenza vaccine had the same subtypes during the two season. Data were analyzed for the 3 subtypes contained in the trivalent vaccine, H1N1, H3N2, B (Yamagata).
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
Participants
  H1N1 | 7 | 7
  H3N2 | 7 | 9
  B (Yamagata) | 7 | 8

3. Secondary Outcome: Number of Adverse Events Definitely or Possibly Related to Vaccination Reported Within 14 Days of Vaccination
Description: Number of adverse events reported within the 14 days after vaccination by each subject within each patient group. Data collected from that reported in safety questionnaires and in Safety Diary that spanned the 14 days post-vaccination.
Time Frame: 0-14 days after vaccination
Population: All adverse events that may have been related are included in this analysis. Events considered not-related were excluded. More information on these AEs is included in the Adverse Events section. All AEs were reviewed by the study DSMB.
Measure: Number; unit: number of AEs reported
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
number of AEs reported
  Local site reaction - grade 1 | 7 | 8
  Local site reaction - grade 2 | 1 | 0
  Other AEs - Grade 1 | 2 | 1

4. Secondary Outcome: Number of Subjects With Seroconversion From T1 to T2 in the High Dose and Standard Dose Vaccine Groups
Description: HAI was measured on blood samples #1 and #2 for all subjects. Seroconversion is defined as a four-fold increase in antibody level between the high-dose and standard-dose recipients within each patient group was performed.
Time Frame: 10-45 days post-vaccination
Population: All participants had blood drawn at baseline (T1) and 10-45 days after vaccination (T2). Analysis was done for the 3 influenza subtypes in the trivalent influenza vaccine. The influenza vaccine was the same in 2013-2014 and 2014-2015.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
Participants
  H1N1 | 3 | 1
  H3N2 | 5 | 5
  B (Yamagata) | 3 | 3

5. Secondary Outcome: Number of Participants Seroprotected at Timepoint 3 in High Dose and Standard Dose Vaccination Groups
Description: Measure HAI on blood sample #3, drawn May-September following vaccination. Report number who still have HAI ≥ 1:40 in the high-dose and standard-dose groups.
Time Frame: at least 5 months post vaccination
Population: Number of subjects seroprotected at T3 for each of the vaccine subtypes. 3 subjects in the HD group and 4 subjects in the SD group were lost-to-follow-up by T3 and not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 4 | 5
Participants
  H1N1 | 4 | 4
  H3N2 | 4 | 5
  B (Yamagata) | 4 | 5

6. Secondary Outcome: Change in Disease Status From Vaccination Through June of the Following Year
Description: Evaluate disease status changes reported by subject on Questionnaire #2 as well as changes reported in clinic notes over the course of the influenza season. Subjects considered "worse" had worsening function of transplanted organ or complications related to underlying condition (e.g. dialysis) or new diagnosis of disease considered serious by PI.
Time Frame: up to 9 months post-vaccination
Population: One subject in the high-dose group was originally on dialysis, but received a kidney transplant during the follow-up period. This subject was excluded from the analysis on change in baseline medical condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 6 | 9
Participants
  Same or better | 5 | 9
  Worse | 1 | 0

7. Secondary Outcome: Number of Adverse Events Considered Definitely or Possibly Related to Vaccination Through Sept 30 of the Year Following Vaccination.
Description: Data gathered from the following
  1. Safety data in 1st 14 days (safety surveys and safety diary)
  2. Safety survey at day 30-45 regarding any unplanned health care visit or other AE during the 30 days after vaccine
  3. On-going passive surveillance of adverse events (AEs)/serious adverse events (SAEs) throughout course of influenza season of enrollment
  4. Chart review of each participant by PI through Sept 30 of the year following vaccine Data collection stopped in September following enrollment.
Time Frame: (1) Date of vaccine through day 30 post-vaccine; (2) Day 31 post-vaccine through September 30 of the year following vaccine
Population: Data used included: active reporting through day 30, survey at end of season, and chart review for data through Sept 30 of the year following vaccination.
Measure: Number; unit: number of AEs reported
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
number of AEs reported
  Day 0 (vaccination) through day 30 | 10 | 9
  Day 31 post-vaccination, through Sept 30 | 0 | 0

8. Other Pre Specified Outcome: Additional Measures of Immunogenicity in High Dose and Standard Dose Vaccinations
Description: This secondary objective was included as exploratory and we plan to add additional analyses when funding is secured. There is no anticipated date when we will have this completed. (No immunogenicity studies have been done besides HAI.) For other immunogenicity: would compare results of blood draw #1 and #2 between the high-dose and standard-dose recipients for each patient group for any of the following: antibody avidity, microneutralization, T-cell interferon, T-cell IL-2, B-cell Immunoglobulin G (IgG) and B-cell Immunoglobulin A (IgA).
Time Frame: 10-45 days post-vaccination
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Numbers of Subjects Who Were Both Seroprotected and Who Seroconverted at T2 and T3 After Vaccination
Description: Seroprotection (HAI>=1:40) and seroconversion (4-fold increase) together have been found to be a better predictor of vaccine effectiveness. Patients had to have both a 4-fold rise in HAI and have HAI>=40 to be counted
Time Frame: (1) T2 measured 14-45 days post-vaccination; (2) T3 measured June 1-Sept 30 post-vaccination (end-of season), following vaccination
Population: For T3, only 4 participants in the high-dose group and 5 participants in the standard-dose group were analyzed due to loss-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
Number analyzed (Participants) | 7 | 9
Participants
  T2 - H1N1 | 3 | 1
  T2 - H3N2 | 5 | 5
  T2 - B (Yamagata) | 3 | 3
  T3 - H1N1: number analyzed (Participants) | 4 | 5
  T3 - H1N1 | 1 | 0
  T3 - H3N2: number analyzed (Participants) | 4 | 5
  T3 - H3N2 | 0 | 1
  T3 - B (Yamagata): number analyzed (Participants) | 4 | 5
  T3 - B (Yamagata) | 1 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from the date of vaccination (T1) through September 30 of the following year. AE data were collected differently over the study. At day 2-7 after vaccination, subjects were called to ask about AEs. Subjects were given a "Diary" to fill out for day 0-14 after vaccination, and the Diary was collected at T2. At day 30-45, subjects were given a questionnaire (in-person at T2 visit or by phone) asking about AEs and any unplanned medical visits during day 0-30 post-vaccine.
Description: In May-June after vaccination, another questionnaire was collected by phone asking about influenza and influenza-like-illness, new health conditions, changes to underlying medical condition, or new immunosuppressive treatments since enrollment. Passive AE data were collected by providing participants with contact information for the study in order to report any concerns.
Arm/Group | Fluzone High Dose | Fluzone Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/9
Other Adverse Events (participants affected / at risk) | 6/7 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone High Dose (N=7) | Fluzone Standard Dose (N=9)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) — Subject developed dialysis catheter insertion site infection 15 days after vaccination. Subject was admitted for IV antibiotics. No long-term sequelae. SAE was determined to be not related to the vaccine by study DSMB.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject developed acute gastroenteritis 27 days after vaccination. Subject required hospitalization for rehydration and monitoring of immunosuppression levels.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone High Dose (N=7) | Fluzone Standard Dose (N=9)
Injection site reaction - pain (General disorders) | 6 (6) | 7 (7) — Pain at site of injection - Grade 1
Injection site reaction - induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Induration at site of injection - Grade 1
Injection site reaction - induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Induration at site of injection - Grade 2
Injection site reaction - bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Bruising at site of injection - Grade 1
Fatigue (General disorders) | 0 (0) | 1 (1) — Fatigue starting a few days after injection - Grade 1, possibly related
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache within 14 days of vaccination - Grade 1, possibly related
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal pain on day after vaccination - Grade 1, possibly related

LIMITATIONS AND CAVEATS:
The number of participants was very low, limiting statistical analysis and limiting the ability to perform any subgroup analysis. Data at T3, were even more limited given loss-to-follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes